CLINICAL TRIAL: NCT04061473
Title: Involvement of Dipeptidyl Peptidase-4 and Sodium-glucose Co-transporter-2 in Extrapancreatic Glucagon Secretion
Acronym: Px-Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Consultant endocrinologist, Professor of Clinical Endocrinology and Director of Center for Clinical Metabolic Research, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-19000992
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Diabetes After Total Pancreatectomy
Keywords: Pancreatectomy; Diabetes; SGLT-2 inhibitor; DPP4 inhibitor; glucagon
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; empagliflozin

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomised, double-blinded, crossover study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pancreatectomized + Placebo (Placebo Comparator): During the experimental day the participant will ingest a standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Before the meal (1 h and 12 h) 1+1 placebo tablets will be administered orally.
  Interventions: Other: Placebo tablet
- Pancreatectomized + DPP-4 inhibitor (Active Comparator): During the experimental day the participant will ingest a standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Before the meal (1 h and 12 h) 1+1 DPP4-inhibitor tablets will be administered orally.
  Interventions: Drug: Sitagliptin 100mg
- Pancreatectomized + SGLT-2 inhibitor (Active Comparator): During the experimental day the participant will ingest a standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Before the meal (1 h and 12 h) 1+1 SGLT-2 tablets will be administred orally.
  Interventions: Drug: Empagliflozin 25 MG
- Healthy + Placebo (Placebo Comparator): During the experimental day the participant will ingest a standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Interventions: Other: Placebo tablet
- Healthy + DPP-4 inhibitor (Active Comparator): During the experimental day the participant will ingest a standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Interventions: Drug: Sitagliptin 100mg
- Healthy + SGLT-2 inhibitor (Active Comparator): During the experimental day the participant will ingest a standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Sitagliptin 100mg — 2 tablets of sitagliptin 100 mg.
  Standardized liquid meal Standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Arms: Healthy + DPP-4 inhibitor; Pancreatectomized + DPP-4 inhibitor
Drug: Empagliflozin 25 MG — 2 tablets of empagliflozin 25 mg.
  Arms: Healthy + SGLT-2 inhibitor; Pancreatectomized + SGLT-2 inhibitor
Other: Placebo tablet — 2 placebo tablets.
  Standardized liquid meal Standardized liquid meal (200 ml) containing: 1,650 KJ, (394 kcal), carbohydrate 50%, protein 15%, fat 35% consisting of glucose (47.2 g + 2.8 g [U-13C6]-glucose), rapeseed oil (14.1 g), whey protein (15.2 g) and 1.5 g paracetamol.
  Arms: Healthy + Placebo; Pancreatectomized + Placebo

SUMMARY:
Glucagon is a 29-amino acid peptide hormone of essential importance for glucose homeostasis. Hitherto glucagon has been believed to be secreted only from the pancreas, but recent studies show that glucagon is also secreted from an extra pancreatic origin - most likely from enteroendocrine cells in the intestinal epithelium (Baekdal et al., unpublished data). This has fundamentally changed the understanding of glucagon physiology and provides new avenues for the investigation of several metabolic disorders in which hyperglucagonaemia represents a common and important pathophysiological characteristic (including type 2 diabetes). To delineate the physiological role of gut-derived glucagon and its potential pathophysiological implications, and thereby clear the way for new treatment modalities targeting gut glucagon, it is of importance to understand how glucagon secretion from the gut is regulated. In contrast to the regulation of pancreatic glucagon secretion, very little is known about the regulation of gut-derived glucagon.

Inhibition of the enzyme dipeptidyl peptidase 4 (DPP-4) which under normal circumstances degrades, and thereby inactivates the two gut-derived incretin hormones, glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide 1 (GLP-1), has been shown to decrease pancreatic glucagon secretion. This is most likely brought about by increased levels of intact, active GLP-1, which is known to suppress pancreatic glucagon secretion. Furthermore, the sodium-glucose transporter 2 (SGLT-2) seems to be implicated in pancreatic glucagon secretion as inhibitors of SGLT-2 have been shown to increase the secretion of pancreatic glucagon secretion.

The present project will employ further investigations of totally pancreatectomised patients to delineate the regulation of gut-derived glucagon secretion with focus on the well-known modulators of pancreatic glucagon secretion, the enzyme DPP-4 and the sodium-glucose co-transporter SGLT-2, respectively.

The study is designed as a randomised, double-blinded, crossover study. 10 healthy persons and 10 totally pancreatectomized patients will be subjected to 3 experimental days. All participants will undergo a screening visit and three experimental days (day A (meal test during DPP-4 inhibition), B (meal test during SGLT-2 inhibition) and C (meal test with placebo)). A liquid meal test will be followed by a fasting period and finished off with an ad libitum meal.

ELIGIBILITY:
Inclusion Criteria:

Pancreatectomised patients

* Caucasian above 30 years of age who have undergone total pancreatectomy
* Blood haemoglobin >7.0 mmol/l for males and >6.5 mmol/l for females
* Informed consent

Non-diabetic control subjects

* Normal fasting plasma glucose and normal HbA1c (according to the World Health Organization (WHO) criteria)
* Normal blood haemoglobin
* Caucasian above 30 years of age
* Informed consent

Exclusion Criteria:

Pancreatectomised patients

* Pancreatectomy within the last 3 months
* Ongoing chemotherapy or chemotherapy within the last 3 months
* Treatment with GLP-1 receptor agonists, DPP-4 inhibitors or SGLT-2 inhibitors within the last 3 months
* eGFR<60 ml/min/1,73m2 and/or albuminuria
* Known liver disease (excluding simple steatosis) and/or serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3 × upper normal limit)
* Pregnancy and/or breastfeeding
* Age above 85 years
* Uncontrolled hypertension and/or significant cardiovascular disease
* Any condition that the investigator feels would interfere with trial participation

Non-diabetic control subjects

* Diabetes or prediabetes (according to WHO criteria)
* First-degree relatives with diabetes
* eGFR<60 ml/min/1,73m2 and/or albuminuria
* Known liver disease (excluding simple steatosis) and/or serum ALAT and/or serum ASAT >3 × upper normal limits)
* Pregnancy and/or breastfeeding
* Age above 85 years
* Uncontrolled hypertension and/or significant cardiovascular disease
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
glucagon excursions measured as incremental area under the curve (iAUC) | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes

SECONDARY OUTCOMES:
PPG excurions measured as incremental area under the curve (iAUC) | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
endogenous glucose production | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
  Using intravenous and oral tracers
GLP-1, gastrin, cholecystokinin, GIP, oxyntomodulin | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
  excurions measured as incremental area under the curve (iAUC)
Differences in gastric emptying, meassurement of s-paracetamol | -120-180 minutes
  measurement of time to peak and incremental area under the curve (iAUC)
satiety, appetite, thirst, | -30, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
  assesed by a visual analougue scale (VAS)
Resting energy expenditure (REE) | -90, 150 and 150 minutes
  measured by indirect calorimetry
p-glucose mmol/L | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
s-peptide pmol/l | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
s-insulin | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
Pulse and blood pressure | -120, -30, -15, 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
  will be measured every 30th min
food intake | 180 and 210 minutes
  the ad libitum meal will be weighed before after ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided